CLINICAL TRIAL: NCT05276154
Title: Clinical Performance of Thermo-Viscous Bulk-Fill Resin Composite Restorations in Comparison to Conventional Bulk-Fill Resin Composite Restorations in Posterior Teeth A Randomized Control Clinical Trial
Brief Title: Clinical Performance of Thermoviscous Bulk Fill Resin Composites in Comparison to Conventional Packable Bulk Fills
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed Amr Kamal, Assistant lecturer (misr university for sciences and technology), Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USPHS for TV bulkfill RC
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thermoviscous bulk fill resin composite (Active Comparator)
  Interventions: Other: thermoviscous bulkfill composite (Viscalor)
- conventional bulk fill resin composite (Active Comparator)
  Interventions: Other: thermoviscous bulkfill composite (Viscalor)

INTERVENTIONS:
Other: thermoviscous bulkfill composite (Viscalor) — a relatively new product of composite resin which is transformed from high viscosity to low viscosity by the action of head produced by a heating device.

SUMMARY:
This clinical trial will be conducted to compare the clinical performance of the thermo-viscous preheated bulk fill composite in the management of carious lesions in posterior teeth in adult patients over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Have at least two molars supported permanent dentition free of any clinically significant occlusal interference and require posterior restoration and fulfilled the inclusion criteria, patients will be informed about the study and will be given an informed consent.

  * The two studied materials restorations should be used in approximately the same sized lesions or within the same extensions.
  * The patient will be reimbursed for attending for the clinical evaluation(s) of their restorations.
  * Be a regular dental attender who agree to return for assessments.

Exclusion Criteria:

* There is history of any adverse reaction to clinical materials of the type to be used in the study.
* There was evidence of occlusal parafunction and/or pathological tooth wear.
* Patients whose history revealed parafunctional habits or use of medications that potentially could cause hyposalivation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
modified United States Public Health Service criteria (USPHS) | 1 year
  scores A,B,C ( A highest score) (C the lowest score) and overall evaluation for the restorations ( Alpha , bravo, charlie, delta) Alpha for the highest score and delta for the lowest scores

SECONDARY OUTCOMES:
post operative senstivity | 1 week

REFERENCES:
- [Background] Balkaya H, Arslan S, Pala K. A randomized, prospective clinical study evaluating effectiveness of a bulk-fill composite resin, a conventional composite resin and a reinforced glass ionomer in Class II cavities: one-year results. J Appl Oral Sci. 2019 Oct 7;27:e20180678. doi: 10.1590/1678-7757-2018-0678. eCollection 2019. PMID 31596369
- [Background] Rickman LJ, Padipatvuthikul P, Chee B. Clinical applications of preheated hybrid resin composite. Br Dent J. 2011 Jul 22;211(2):63-7. doi: 10.1038/sj.bdj.2011.571. PMID 21779058
- [Background] Wagner WC, Aksu MN, Neme AM, Linger JB, Pink FE, Walker S. Effect of pre-heating resin composite on restoration microleakage. Oper Dent. 2008 Jan-Feb;33(1):72-8. doi: 10.2341/07-41. PMID 18335736
- [Background] Rueggeberg FA, Daronch M, Browning WD, DE Goes MF. In vivo temperature measurement: tooth preparation and restoration with preheated resin composite. J Esthet Restor Dent. 2010 Oct;22(5):314-22. doi: 10.1111/j.1708-8240.2010.00358.x. PMID 21029335
- [Background] Costa T, Rezende M, Sakamoto A, Bittencourt B, Dalzochio P, Loguercio AD, Reis A. Influence of Adhesive Type and Placement Technique on Postoperative Sensitivity in Posterior Composite Restorations. Oper Dent. 2017 Mar/Apr;42(2):143-154. doi: 10.2341/16-010-C. Epub 2016 Nov 28. PMID 27892839
- [Background] Campbell I, Kang J, Hyde TP. Randomized Controlled Trial of Postoperative Sensitivity with Warm and Room Temperature Composite. JDR Clin Trans Res. 2017 Jul;2(3):295-303. doi: 10.1177/2380084416682934. Epub 2016 Dec 20. PMID 30938633
- [Background] Lempel E, Ori Z, Szalma J, Lovasz BV, Kiss A, Toth A, Kunsagi-Mate S. Effect of exposure time and pre-heating on the conversion degree of conventional, bulk-fill, fiber reinforced and polyacid-modified resin composites. Dent Mater. 2019 Feb;35(2):217-228. doi: 10.1016/j.dental.2018.11.017. Epub 2018 Nov 28. PMID 30503020
- [Background] Demirel G, Orhan AI, Irmak O, Aydin F, Buyuksungur A, Bilecenoglu B, Orhan K. Micro-computed tomographic evaluation of the effects of pre-heating and sonic delivery on the internal void formation of bulk-fill composites. Dent Mater J. 2021 Mar 31;40(2):525-531. doi: 10.4012/dmj.2020-071. Epub 2020 Dec 2. PMID 33268693
- [Background] Loumprinis N, Maier E, Belli R, Petschelt A, Eliades G, Lohbauer U. Viscosity and stickiness of dental resin composites at elevated temperatures. Dent Mater. 2021 Mar;37(3):413-422. doi: 10.1016/j.dental.2020.11.024. Epub 2021 Jan 19. PMID 33353736
- [Background] Yang J, Silikas N, Watts DC. Pre-heating time and exposure duration: Effects on post-irradiation properties of a thermo-viscous resin-composite. Dent Mater. 2020 Jun;36(6):787-793. doi: 10.1016/j.dental.2020.03.025. Epub 2020 May 5. PMID 32386715
- [Background] Marcondes RL, Lima VP, Barbon FJ, Isolan CP, Carvalho MA, Salvador MV, Lima AF, Moraes RR. Viscosity and thermal kinetics of 10 preheated restorative resin composites and effect of ultrasound energy on film thickness. Dent Mater. 2020 Oct;36(10):1356-1364. doi: 10.1016/j.dental.2020.08.004. Epub 2020 Sep 1. PMID 32888725
- [Background] Ebrahimi-Chaharom ME, Safyari L, Safarvand H, Jafari-Navimipour E, Alizadeh-Oskoee P, Ajami AA, Abed-Kahnamouei M, Bahari M. The effect of pre-heating on monomer elution from bulk-fill resin composites. J Clin Exp Dent. 2020 Sep 1;12(9):e813-e820. doi: 10.4317/jced.56989. eCollection 2020 Sep. PMID 32994869
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/32446504/